CLINICAL TRIAL: NCT00334191
Title: A Randomised, Double Blind, Placebo Controlled Pilot Study of the Effect of Sodium Bicarbonate on Postoperative Renal Function and Oxidative Stress in Patients Undergoing Elective Cardiopulmonary Bypass.
Brief Title: Sodium Bicarbonate in Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H2005/02249
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Cardiac Surgery and Cardiopulmonary Bypass
Keywords: Cardiac surgery,; Cardiopulmonary bypass,; Oxidative stress,; Acute renal dysfunction,; Sodium Bicarbonate
MeSH Terms: interventions — Sodium Bicarbonate

INTERVENTIONS:
Drug: Sodium Bicarbonate
Drug: Placebo

SUMMARY:
Many patients develop kidney failure after cardiac surgery. Although this kidney failure can usually be treated effectively, a longer stay in intensive care is often required. While many patients suffer no long term ill effects after developing post-operative kidney failure, some require long term kidney dialysis. We also know that patients who develop post-operative kidney failure are much more likely to die before they leave hospital.

Why some people develop kidney failure after cardiac surgery is not known. However, doctors suspect that the process of cardiopulmonary bypass (where the functions of the heart and lungs are taken over by a machine during the operation, to allow the surgeon to operate) overactivates some of the same mechanisms the body uses to defend itself against severe infection.

Many of the cell changes by which severe infection causes kidney failure also occur after cardiopulmonary bypass. One of the main overactive defence mechanisms is the release of highly toxic compounds derived from oxygen - a process called 'oxidative stress'.

The investigators believe that sodium bicarbonate might reduce the oxidative stress, which occurs during cardiac surgery, and so prevent or decrease the kidney failure, which occurs in many patients.

The investigators hope to give sodium bicarbonate (in similar doses to those used safely for treatment of acidosis) to patients during, and for 24 hours after cardiac surgery, and to compare the effects with patients who have not had sodium bicarbonate. The drug, or a placebo, will be given through the drip, which is present in all cardiac surgery patients. Whether a particular patient receives the drug or placebo will be decided at random, and neither the patient nor the investigators will know which has been given. We will measure kidney function before and after the operation using the standard blood tests.

The investigators will also take four 20ml samples of blood, spaced before, during, and after the operation, from the arterial catheter routinely inserted in every patient. This blood would be used to measure oxidative stress, and also some of the proteins inside the blood cells, which are responsible for creating the toxic oxygen compounds. In this way we will discover not only the effect of sodium bicarbonate, but also the mechanism of that effect.

Sodium bicarbonate is commonly used to treat metabolic acidosis in severe renal disease, circulatory insufficiency due to shock or severe dehydration and has been shown to be an effective drug in preventing contrast-induced nephropathy.

Sodium bicarbonate is considered to be safe in the setting of intensive care treatment and is often used in the treatment of patients with metabolic acidosis without any discernible adverse clinical effects.

This is a pilot study. If the drug proves effective in this context, further studies on a larger scale would be required to justify its general use.

There will be no extra risk to a patient who participates in the study, and no discomfort other than that normally associated with cardiac surgery.

Informed consent will be obtained from the patient prior to the operation by one of the investigators or the ICU research nurse. The clinical care of a patient who does not consent for any reason will not be affected.

DETAILED DESCRIPTION:
Renal impairment following cardiopulmonary bypass is common. 11.4% to 42% of patients with previously normal renal function show a postoperative rise in serum creatinine. While most of these patients do not require either short or long term renal replacement, the mortality of patients with acute renal failure is substantially greater than those who do not develop renal dysfunction1.

Cardiopulmonary bypass activates components of the non-specific immune system, which leads to the generation of compounds containing oxygen free radicals. A study of 14 patients undergoing cardiac surgery found increased levels of serum lipid peroxidation products (thiobarbituric acid reactive substances) within 15 minutes of the commencement of cardiopulmonary bypass, which returned to preoperative levels by the following morning. The total serum antioxidative capacity was correspondingly decreased intraoperatively, and remained decreased at 24 hours postoperatively. A similar study of total plasma antioxidant status showed decreased levels up to 72 hours postoperatively. It is clear that cardiopulmonary bypass causes oxidative stress and depletion of antioxidant capacity.

N-Nitrosation of oxygenated nitric oxide (NO.) solutions was previously shown to be significantly inhibited by the strong scavenging ability of NaBic presumably by anion scavenging of nitrosating agents. At physiologic concentrations, NaBic scavenges peroxynitrite and reactive oxygen species generated from nitric oxide. This may contribute to a reduction in the deleterious effects of NO generating agents. NaBic is therefore a potential regulator of NO-induced toxicity. NaBic is considered to be safe in the setting of intensive care treatment and is often used in the treatment of patients with metabolic acidosis without any discernible adverse clinical effects. NaBic increases the pH-level by buffering of hydrogen ions, which can cause electrolyte balance shifts, e.g. Potassium will be shifted increasingly intracellular. Frequent control of pH and potassium levels is required to prevent alkalosis and hypokalemia. These adverse effects are uncommon or typically only biochemical in nature.

Oxidative stress can be produced experimentally using hypertonic glycerol. Intramuscular injection of hypertonic glycerol in rats precipitates acute renal failure associated with a marked decrease in renal reduced levels of antioxidative agents. Pre-treatment with NaBic is more protective than sodium chloride in animal models of acute renal failure secondary to ischaemia or doxorubicin.

Radio-contrast dye commonly causes renal dysfunction, in part through oxidative stress in the kidney. While not an approved indication, intravenous sodium bicarbonate has been used successfully to attenuate radiocontrast-induced nephropathy, and was more effective than standard intravenous fluid prophylaxis. Hydration with NaBic before contrast exposure is more effective than hydration with sodium chloride for prophylaxis of contrast-induced renal failure. By increasing medullary pH in the kidneys, NaBic might protect from oxygen injury by slowing pH-dependent radical production.

While never investigated for its effects on renal function after cardiac surgery, the effect of perioperative sodium bicarbonate on other systems has been studied.

In a clinical trial with 15 infants who were mechanically ventilated during the immediate postoperative period after corrective cardiac surgery sodium bicarbonate increased the arterial pH, lowered the mean pulmonary arterial pressure and increased the cardiac index resulting in a decrease in pulmonary vascular resistance. Infusion of sodium bicarbonate resulted in a significant improvement in skin microcirculatory perfusion in an observation study with 15 patients undergoing cardiopulmonary bypass.

The negative effects of peroxynitrite causing oxidative stress after tyrosine nitration in neurodegenerative disorders were strongly reduced in the presence of sodium bicarbonate in in-vitro experiments.

There is thus evidence that sodium bicarbonate affects the cardiovascular, respiratory and immune systems and may be of benefit to patients undergoing cardiac surgery.

Hypotheses Sodium bicarbonate administered from the time of induction of anaesthesia prior to cardiac surgery and for 24 hours postoperatively results in a decreased change in renal function measured as serum creatinine change greater than 25% from baseline to peak level within first five postoperative days.

Secondary outcomes which will be measured include:

* change in serum creatinine greater than 50% from baseline to peak level

  . creatinine clearance over the first postoperative day;
* length of ventilation;
* ICU stay;
* hospital stay;
* serum creatinine levels on day 2 post-op;
* plasma antioxidant activity;
* NF-kB activation in the cellular components of blood;
* pro-inflammatory cytokine response
* Activation of the nitric oxide synthase pathway

Study Design - overview and rationale

Patients will be randomised to receive sodium bicarbonate in 5% dextrose from the induction of anaesthesia until 24 hours postoperatively, or a placebo (vehicle) (154mEq/L saline in 5% dextrose solution).

Serum creatinine is the most commonly used clinical indicator of renal function along with urine output. Both will be measured for 48 hours postoperatively - the time period during which renal impairment is most likely to develop. A more sensitive indicator of renal dysfunction is creatinine clearance. This will be measured over the first 24 hours postoperatively.

The efficacy of sodium bicarbonate in preventing oxidative stress will be assessed using a measure of total plasma antioxidant activity (the bathocuproine assay) and by quantification of the 8-isoprostane levels.

Any renal effect of sodium bicarbonate will be correlated with levels of plasma pro-inflammatory cytokines (IL-1, IL-6 and TNF-alpha), which are known to be associated with oxidative-stress induced renal failure. Activation of inducible nitric oxide production is also associated with renal failure, and the effect of sodium bicarbonate on nitric oxide synthase mRNA expression in the cellular components of blood will be assayed by real-time PCR. Nitric oxide production will be assessed by measurement of plasma nitrotyrosine concentration. Assay of nitrotyrosine is superior to the traditional Greiss reaction (which measures nitrate and nitrite derivatives of nitric oxide), as nitrate and nitrite undergo renal excretion, and many of these patients will have altered renal function.

At a molecular level, many of the genes responsible for stimulating oxidative stress are regulated by the promoter NF-kB. The cellular components of blood will be assayed for NF-kB using an established ELISA technique. NF-kB in the cellular components of blood will also be assayed using real-time PCR.

Randomisation

The randomisation will be based on random numbers generated by computer. Once consent is obtained, the allocation of either treatment with Sodium Bicarbonate or placebo will be organised by an independent person (clinical trials pharmacist) who will dispense the coded infusion bags. This will be delivered to the anaesthetic staff looking after the patient in theatre, and the ICU nurse caring for the patient postoperatively.

Detailed protocol

Immediately following the induction of anaesthesia, prior to the first surgical incision, Sodium Bicarbonate will be administered in a dose of 154mEq/L in 5% dextrose over 60 mins (3mL/kg/h) followed by continuous IV infusion of 154mEq/L in 5% dextrose over 23 hours (1mL/kg/h) or placebo (154mEq/L saline in 5% dextrose). Patients randomised to receive placebo will receive an equivalent volume of dextrose. The appearance of the dextrose solution and sodium bicarbonate solutions is similar, and there will be no marking on the infusion bag other than an identifying study number.

A 24 hour urine collection will begin immediately on arrival in ICU, to allow determination of creatinine clearance. This will be measured in the hospital clinical pathology laboratory.

Clinical data will be recorded as detailed below by the investigators or the ICU research nurse.

20 ml samples of heparinized blood will be taken from the arterial line for cytokine and molecular analysis. Samples will be taken immediately after the induction of anaesthesia, on arrival in the intensive care unit, and 6, 12 and 24 and 72 hours postoperatively. Immediately following collection, the blood will be centrifuged at low speed to separate the plasma from the cellular components, both of which will be stored in aliquots at -70 degrees prior to batch analysis.

Analysis of plasma total antioxidant activity and 8-isoprostane, IL-1, IL-6, TNF-alpha and nitrotyrosine concentrations will be performed using commercially available ELISA reagent kits (Oxford Biomedical Research, Oxis Research, BioCore). The cellular components of blood will be assayed for NF-kB concentration using a commercially available ELISA kit (Oxford Biomedical Research), also for iNOS and NF-kB mRNAs using a real-time PCR machine and Applied Biosystems pre-developed assay reagents with 18S as the endogenous control. The principal investigator has experience of these or similar techniques.

Statistics and power calculation Using data available from our cardiac surgery database of over 2500 patients in the last 5 years, we expect 50% of patients developing an increase in serum creatinine greater than 25% from baseline to peak in the control group.

Given a minimal clinically important reduction of this proportion to 30% in the Sodium Bicarbonate group, 100 patients are needed to have a 90% power of detecting a difference between the control and the intervention group at an alpha of 0.05.

Data collection Data collection will be performed by the principal investigator, ICU research nurse and ICU nursing staff.

The following variables will be obtained:

Code for patient, gender and age. Date of admission to ICU Operative procedure and time on cardiopulmonary bypass Preoperative assessment of left ventricular function Serum creatinine and urea preoperatively, immediately postoperatively, 12 and every 24 hours thereafter (as measured for clinical purposes). Doses of frusemide administered (or rate of frusemide infusion) Use of inotropes Cardiac output whenever measured for clinical purposes in the first 24 hours postoperatively Urine output in each 6 hour period for the 24 hours postoperatively Date of discharge from ICU and hospital or death

Resources required The principle of the study has been discussed with the involved cardiac anaesthetists, cardiac surgeons, intensivists and intensive care nurses, who have offered their co-operation. ICU research nurse to allocate patients and collect clinical data. Pharmacy will be required to prepare drug and placebo infusion bags. Clinical pathology will be required to perform 24 hour creatinine clearance estimation (in addition to those tests clinically indicated)

Protocol violations All protocol violations will be recorded. It will then be decided whether the nature of such violation had been such that the patient should be excluded from primary data analysis. Such evaluation will be blinded to treatment.

Withdrawal The treating clinician will have the right to withdraw the patient from the study if he or she believes that continued participation is jeopardising the patient's well being.

Ethical Issues Sodium bicarbonate used in this study is considered to be very safe as has been demonstrated by its widespread clinical use in the management of critically ill patients with metabolic acidosis. We consider the potential benefit of this treatment theoretically significant. Given the balance of benefits and risks, the investigators consider it ethical to proceed and seek informed consent.

Indemnity This is an investigator-initiated study and, accordingly, no commercial sponsor's indemnity has been provided.

ELIGIBILITY:
Inclusion Criteria:

* Age above 70 years
* Preexisting renal impairment (preoperative serum creatinine level >120µmol/L
* New York Heart Association class III/IV or Moderate to poor left ventricular dysfunction
* Valve surgery or complex cardiac surgery
* Redo cardiac surgery
* Insulin-dependent diabetes mellitus

Exclusion Criteria:

* Age <18 years
* Emergency cardiac surgery
* Planned off-pump cardiac surgery
* Enrolled in conflicting research study
* Known blood-borne infectious disease
* Chronic inflammatory disease on immunosuppression
* Chronic moderate to high dose corticosteroid therapy (>10mg/d prednisone or equivalent)
* End stage renal disease (serum creatinine >300µmol/L)
* Thiamine deficiency will be excluded on medical and dietary history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Proportion of patients developing an increase in serum creatinine greater than 25% from baseline to peak level within first five postoperative days.

SECONDARY OUTCOMES:
Proportion of patients developing an increase in serum creatinine greater than 50% from baseline to peak level within first five postoperative days.
Relative change in serum creatinine,
Urinary output,
Use of renal replacement therapy (RRT),
Acute renal dysfunction,
Duration of ventilation,
Chest tube drainage,
Need for return to operating room,
Incidence of post-operative atrial fibrillation (AF),
Duration of stay in the intensive care unit (ICU)
Duration of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MD, FRACP, Principal Investigator — Austin Health
Locations (1):
- Austin Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Haase M, Haase-Fielitz A, Bellomo R, Devarajan P, Story D, Matalanis G, Reade MC, Bagshaw SM, Seevanayagam N, Seevanayagam S, Doolan L, Buxton B, Dragun D. Sodium bicarbonate to prevent increases in serum creatinine after cardiac surgery: a pilot double-blind, randomized controlled trial. Crit Care Med. 2009 Jan;37(1):39-47. doi: 10.1097/CCM.0b013e318193216f. PMID 19112278
- [Derived] Haase M, Haase-Fielitz A, Ratnaike S, Reade MC, Bagshaw SM, Morgera S, Dragun D, Bellomo R. N-Acetylcysteine does not artifactually lower plasma creatinine concentration. Nephrol Dial Transplant. 2008 May;23(5):1581-7. doi: 10.1093/ndt/gfm818. Epub 2008 Jan 17. PMID 18202091